CLINICAL TRIAL: NCT05361876
Title: Remote Sensing and Measurements of Hemodynamic Changes in Blood Flow for Wingate Anaerobic Test Using a Novel Image Processing Algorithm.
Brief Title: Thermographic Analysis of Hemodynamics Changes Through & Following Wingate Test
Status: Completed | Type: Observational
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Mickey Scheinowitz, PhD, Professor, PhD FACSM, Tel Aviv University
Other Study IDs: TAU BioMed 123456
Record Dates: First submitted 2022-04-25; First posted 2022-05-05 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Health, Subjective

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young Male: Healthy men with some sport experience
- Young Female: Healthy female with some sport experience

SUMMARY:
Remote sensing and measurements of hemodynamic changes in blood flow for Wingate Anaerobic test using a novel image processing algorithm. The algorithm calculates the heat distribution from the thermal images and assesses the changes in blood flow and temperatures in the torso and legs for each individual participant.

DETAILED DESCRIPTION:
Remote sensing and measurements of hemodynamic changes in blood flow during and following the Wingate Anaerobic test using Infra-Red (IR) cameras with novel image processing algorithms. The algorithm calculates the heat distribution from the thermal images and computes the changes in temperatures measured in the torso and that measured in the lower limbs before the test, immediately after, and during 10 minutes recovery period.

Background Thermal imaging The human body is self-generating and regulates the essential levels of temperature for survival. The body core is relatively stable in temperature, but the shell of the body (the surface tissues, which are mainly the skin) forms part of the regulatory process. Body temperature has been used to study many diseases where skin temperature can depict the presence of inﬂamation in underlying tissues, or where blood ﬂow is increased or decreased because of a clinical abnormality. Thermal imaging has been investigated for numerous medical applications. Several studies reviewed medical thermography [1-3]. Thermal imaging has been investigated for bowel ischemia [4], fever screening [5], diabetic foot, vascular disorder [6], thermoregulation study [7], and breast cancer [8].

Wingate Test In the last 50 years, the Wingate Test is considered to be a common standard for the assessment of the anaerobic capability of athletes. The test is usually performed on computerized stationary bikes, while the participant has to pedal as hard as possible for only 30 seconds at resistance equivalent to 0.075 of their body weights (3).

A previous study (4) has shown a high correlation between the effective power generated and the hemodynamic changes between the leg muscles and the thoracic area of the participant.

Acute hemodynamic changes are the result of intensive vasodilation of metarterioles surrounding the main leg muscles and heavy blood perfusion. The massive blood flow in these areas causes congestion and slows the venous return to the heart.

During this phase, we expect to see significant temperature change between the warm legs, and relatively cooler heart (torso). As the recovery phase progress, we expect to see the legs cool down and the torso warms up until homeostasis is reached.

Thermal imaging and analysis The thermal imaging analysis will be performed using MATLAB software to extract two main features: mean temperature and the entropy, in a selected region-of-interest (ROI). First, the thermal image parameters will be stored in an EXCEL file as a two-dimensional matrix of temperature values. Then, the image (CSV file) is read to the program and the entire matrix is divided into the maximal temperature in the image. This yields a set of normalized temperatures in which the maximal value is 1 and which will be measured at rest, before the Wingate test has been performed. (This normalization is required to obtain correct entropy values using the MATLAB command.) The image is then resized fourfold in each axis and the result is displayed to the user. The user manually selects from this image a rectangular region, and the program extracts the mean value and the entropy of this region. The obtained mean value is multiplied by the maximal temperature in the original image (before normalization) to get the actual mean temperature (rather than the normalized temperature) in the selected ROI.

The main study goal suggests a correlation between the power generated during the 30 seconds of the Wingate Test and the temperature difference between the hot legs and relatively cold torso.

Method: 16 - 20 participants (10 men + 10 Women) healthy, age: 18-38, with some sports experience.

Candidates will be screened by questionnaire + verbal interview, and then they'll sign the Voluntary Informed Consent form (copy attached). Each participant will do his test alone for about one hour.

Test procedure: 5 minutes of warm-up, 2 minutes rest, ½ minute test, 10-15 minutes staying relaxed on the bike while the IR cameras are taking photographs synchronously every minute.

Data gathering: 3 IR cameras (ONE Pro) will be fixed on 3 tripods, one for each leg, and one for the torso photographing. A Voice recorder will record every individual test completely.

Data analysis The picture analysis will provide us with average (right & left) legs and torso temperatures every minute from test start and 15 minutes later.

The SRM® bike computer will produce a power graph over 30 seconds of the test + Heart Rate recording of the participant for 15 minutes.

Assuming a positive correlation between the average output power, and the temperature difference (legs vs torso), we'll draw a graph of all participants.

Additional outcome results: Time required to full recovery - homeostasis, Heart Rate (HR) changes during recovery time. We may compare these additional results to the main correlation graph.

ELIGIBILITY:
Inclusion criteria:

* Age 18 up to 38 years old
* Good health record
* Sports experience of minimum 2 years

Exclusion criteria:

* Recorded health issues
* Sedentary type people

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Israeli volunteers
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Temperatures of face, torso and legs, during and following Wingate Tests | 30 minutes
  The calculated skin area temperatures, following the sensing and measurements of temperature changes during and following the Wingate Anaerobic Test, using a novel image processing algorithm. The algorithm calculates the heat distribution from the thermal images and assesses the temperature changes in the face, torso, and legs of each individual participant.

SECONDARY OUTCOMES:
Participant's maximum anaerobic legs power on SRM® bicycles | 30 seconds
  This specific Wingate test is performed on SRM® stationary bicycles. SRM computer adjusts the bicycle's resistance to match the maximum capability of the participant while measuring and recording the applied power in watts, over a period of 30 seconds.
Time required to full recovery - homeostasis | 10 - 15 minutes
  Measuring the time from test end, until hemodynamics homeostasis returns

CONTACTS AND LOCATIONS:
Overall Officials: Mickey Schenowitz, Prop. FACSM, Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, POBox 39040,, Israel

IPD SHARING:
Plan to Share IPD: Yes
Coded list for all participants. Data per participant will include: Performed power, Heart rate, body temperature map
Supporting Information: Study Protocol, ICF, CSR
Time Frame: During all tests effective time, current - until December 31st, 2021
Access Criteria: Coded details, as a part for a planned medical article